## The Feasibility of Engage Therapy With Video Support for Homebound Older Adults

Clinical trials number: NCT05346055

## **Primary investigator:**

Natalie C. Benda, PhD 560 West 168th Street, New York, NY 10032 Room 623 212-305-9547 nb3115@cumc.columbia.edu

## Sponsor:

Weill Cornell Medical College of Cornell University

## Statistical analysis plan

We had planned to analyze baseline, interim, and post-study assessment data will be analyzed using statistical hypothesis testing with appropriate parametric or non-parametric tests as dictated by the nature of the assessment output and the distribution of the data collected. Given our resultant study sample with a small N of completed subjects, data will be analyzed simply using descriptive statistics (e.g., mean, standard deviation).